CLINICAL TRIAL: NCT03663127
Title: Evaluation of "Beauty Drink" on Regulation of Blood Pressure Effect by Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, You-Cheng Shen, Associate Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CS18077
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Hypertension
Keywords: gamma-aminobutyric acid; blood pressure; clinical trial; angiotensin converting enzyme; Beauty Drink
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beauty Drink (Experimental): Subjects receive two bottles "Beauty Drink" per day for 8 weeks of a stage.
  Interventions: Dietary Supplement: Beauty Drink
- Placebo (Placebo Comparator): Subjects receive two bottles placebo per day for 8 weeks of a stage.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beauty Drink — Subjects receive two bottles of "Beauty Drink" per day for 8 weeks of a stage. Anthropometric measurements such as blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]), body weight, body fat, waistline, hips, and blood biochemical parameters including FBG, albumin, TC, TG, HDL-C, LDL-C, Cr, BUN, AST, and ALT were measured every four weeks.
  Arms: Beauty Drink
Dietary Supplement: Placebo — Subjects receive two bottles of placebo of similar appearance per day for 8 weeks of a stage. In addition, anthropometric measurements such as blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]), body weight, body fat, waistline, hips, and blood biochemical parameters including FBG, albumin, TC, TG, HDL-C, LDL-C, Cr, BUN, AST, and ALT were measured every four weeks.
  Arms: Placebo

SUMMARY:
This report assesses the effect of supplementation with gamma-aminobutyric acid on blood pressure among people with mild hypertension. Overall, "Beauty Drink" consumption for 8 weeks could successfully reduce mean diastolic and systolic BP through the suppression of ACE linked to downstream suppression of angiotensin II formation, which further decreases the sympathetic outflow leads to hypertension.

DETAILED DESCRIPTION:
This report assesses the effect of supplementation with gamma-aminobutyric acid on blood pressure among people with mild hypertension. Fifty subjects with systolic blood pressure (SBP) between 120 and 159 mm Hg and/or diastolic blood pressure (DBP) between 80 and 99 mm Hg were randomized to ingest 2 bottles of "Beauty Drink" or placebo per day for 8 weeks of a stage. In addition, anthropometric measurements (blood pressure, body weight, body fat) and blood biochemical markers including fasting blood glucose (FBG), albumin, total cholesterol (TC), triglyceride (TG), HDL-C, LDL-C, creatinine (Cr), blood urea nitrogen (BUN), AST, ALT were examined every four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects were untreated hypertensive men or women aged between 20 and 70 years old with SBP between 120 and 159 mmHg and/or DBP between 80 and 99 mmHg as measured in a sitting position

Exclusion Criteria:

* Subjects were excluded if they had a history of major cardiovascular disease or severe liver dysfunction; Diastolic blood pressure ≥ 100 mmHg or Systolic blood pressure ≥ 160 mmHg;
* Alcoholic;
* US-controlled diabetics;
* Stoke in past one year;
* Mental diseases or melancholia;
* Pregnancy or breast-feeding a child;
* Renal dysfunction;

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
The changes of blood pressure of the subjects (SBP and DBP) | 8 weeks
  values change of systolic and diastolic BPs between before to after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: You-Cheng Mr Shen, Ph.D., Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan